CLINICAL TRIAL: NCT00680979
Title: Preventing Excessive Weight Gain in Adolescent Girls at High-Risk for Adult Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080139; 08-CH-0139
Record Dates: First submitted 2008-05-17; First posted 2008-05-20 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2015-08-20

CONDITIONS: Obesity; Overweight; Binge Eating
Keywords: Prevention; Obesity; Binge Eating; Adolescents; Overweight; Weight Gain
MeSH Terms: conditions — Obesity; Overweight; Bulimia; Weight Gain | interventions — Interpersonal Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy
Behavioral: Health Education

SUMMARY:
This study will examine whether interpersonal psychotherapy (IPT) can help reduce excessive weight gain in adolescent girls. It will compare the effectiveness of IPT with a teen health education program in preventing weight gain.

Adolescent girls between 12 and 17 years of age who are at risk for becoming overweight adults, by virtue of being above average weight and experiencing episodes of loss of control over eating, may be eligible for this study. Candidates are screened in two visits with the following procedures:

Visit 1

* Height and weight measurements.
* Interview and questionnaires about the child s general health, social and psychological functioning and eating patterns and behaviors.

Visit 2

* Physical examination, blood and urine tests.
* DXA scan to measure body fat, muscle and bone mineral content.
* Laboratory test meal. The child fills out a rating scale about her level of hunger and is then given a food buffet from which she is instructed to eat as much as she wants. Immediately after eating, the child again completes the hunger rating forms.
* Interview about the child s mood and psychological functioning.

Participants are assigned at random to either the IPT or teen health education program. All participants have a 1- to 1 1/2-hour individual session with a therapist, followed by 12 weekly group sessions of 1 1/2 hours each in their assigned program. They are assessed at the end of the program with questionnaires and body measurements. They return to the clinic after 6 months for body measurements, blood test, DXA scan, questionnaires, interview and a test meal, and again at 1 year for body measurements, questionnaires and a DXA scan.

DETAILED DESCRIPTION:
The most prevalent disordered eating pattern described in overweight youth is loss of control (LOC) eating, during which individuals experience an inability to control the amount of food they are consuming. LOC eating appears to be associated cross-sectionally with greater adiposity in children and adolescents, and appears to predispose youth to gain weight or body fat above that expected due to normal growth, thus likely contributing to obesity in susceptible individuals. Interpersonal Psychotherapy (IPT), a form of psychotherapy that has been adapted for the treatment of eating disorders, has demonstrated efficacy in reducing binge eating episodes and inducing modest weight loss (or at least weight stabilization) among adults diagnosed with binge eating disorder. We adapted group IPT for the targeted prevention of excessive weight gain (IPT-WG) among adolescent girls. Our pilot data support the feasibility and acceptability of a 12-week group IPT-WG trial among adolescent girls at high risk for obesity who report LOC eating, and preliminary findings suggest that IPT-WG has the potential to prevent excessive weight gain. We now propose an adequately powered clinical trial to evaluate the efficacy of IPT-WG compared to a standard-of-care health education for stabilizing weight and body fat gain trajectories in 117 adolescent girls at high risk for adult obesity who report LOC eating. Participants will be randomly assigned to a 12-week group IPT-WG or health education group; anthropometric variables will be measured at baseline, immediately after, and for up to 1 year following the initiation of treatment. We will assess the efficacy of IPT-WG in improving social functioning and reducing negative mood, disturbed eating patterns, and emotional distress. We also aim to determine the impact of IPT-WG on objective measures of LOC eating during a test meal and on appetitive hormones.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria.

* Female.
* Age 12 17 years.
* BMI between 75th and 97th percentile.
* English speaking.
* Good general health.
* Participants must have normal laboratory testing, including negative urine glucose and normal electrolytes, hepatic, and thyroid function, or they will be referred for treatment.

EXCLUSION CRITERIA:

Individuals will be excluded (and referred to non-experimental treatment programs as needed):

* Presence of major illnesses: renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication). Non-serious medical illnesses, such as seasonal allergies, will be reviewed on a case-by-case basis.
* Presence of an obesity-related medical complication that would require a more aggressive weight loss intervention approach. Such comorbidities include hyperlipidemia (LDL-cholesterol greater than 160 mg/dL), hypertension (defined by age-, sex-, and height- specific standards fasting hyperglycemia (fasting glucose greater than 100 mg/dL) and nonalcoholic steatohepatitis (ALT above NIH Clinical Center laboratory norms with consistent radiologic findings and absence of another cause such as infectious hepatitis).
* Regular use of prescription medications. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study. Individuals taking medications for most conditions will be excluded, but medication use for non-serious conditions (e.g., acne) will be considered on a case-by-case basis. In particular, participants currently prescribed SSRIs, neuroleptics, tricyclics, stimulants, or any medication known to affect body weight or eating will be excluded.
* Current involvement in psychotherapy or a structured weight loss program.
* Weight loss during the past 2 months for any reason exceeding 3 per cent of body weight.
* Pregnant or recently pregnant girls (within 1 year of delivery).
* History of an eating disorder or a current eating disorder (other than binge eating disorder) as determined by medical history or if uncovered during the study s structured clinical interviews. Subjects found to have an eating disorder other than binge eating disorder at baseline will be referred to mental health specialists for further evaluation and treatment.
* Current pregnancy or breast feeding. A negative pregnancy test before starting the study will be required. Because pregnancy is a state in which weight gain is expected and appropriate, pregnant individuals would not be suitable for this study. Sexually active females must be using an effective form of birth control. These methods include total abstinence (no sex), oral contraceptives ( the pill ), an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended. Should a participant in the IPT-WG group become pregnant during the 12 weeks of therapy, she will be excluded from the group sessions. The girl s IPT-WG therapists will closely assist her in obtaining an appropriate referral to a community mental healthcare provider. The IPT-WG leaders will request a release of information so that they may communicate with the community therapist in order to facilitate a smooth transition for the girl.
* Individuals who have DSM-IV-TR major depressive disorder, psychoses, current substance or alcohol abuse, conduct disorder, or a diagnosed psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study. Individuals whose parents or guardians have current substance abuse or a diagnosed psychiatric disorder or other condition that, in the opinion of the investigators, would impede adherence with the study.
* Inability to participate in a group due to psychiatric or cognitive functioning. School placement (e.g. grade level) will be used as an estimate of cognitive functioning. The decision to include or exclude subjects for this reason is left entirely to the discretion of the investigators.
* Any other condition in the adolescent or her parents or guardians that, in the opinion of the investigators, would impede compliance or possibly hinder completion of the study.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2008-05-15; Primary Completion 2015-04-16 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Girls with LOC eating will be randomly assigned to IPT-WG or HE to examine their expected BMI change based upon CDC BMI growth chart data versus their actual in BMI over the course of two years. | 1 year

SECONDARY OUTCOMES:
Efficacy of IPT-WG in improving socia | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - United States Uniformed Health Service, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Ogden CL, Kuczmarski RJ, Flegal KM, Mei Z, Guo S, Wei R, Grummer-Strawn LM, Curtin LR, Roche AF, Johnson CL. Centers for Disease Control and Prevention 2000 growth charts for the United States: improvements to the 1977 National Center for Health Statistics version. Pediatrics. 2002 Jan;109(1):45-60. doi: 10.1542/peds.109.1.45. PMID 11773541
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Derived] Shank LM, Tanofsky-Kraff M, Radin RM, Shomaker LB, Wilfley DE, Young JF, Brady S, Olsen CH, Reynolds JC, Yanovski JA. Remission of loss of control eating and changes in components of the metabolic syndrome. Int J Eat Disord. 2018 Jun;51(6):565-573. doi: 10.1002/eat.22866. Epub 2018 Apr 1. PMID 29607525
- [Derived] Tanofsky-Kraff M, Shomaker LB, Wilfley DE, Young JF, Sbrocco T, Stephens M, Brady SM, Galescu O, Demidowich A, Olsen CH, Kozlosky M, Reynolds JC, Yanovski JA. Excess weight gain prevention in adolescents: Three-year outcome following a randomized controlled trial. J Consult Clin Psychol. 2017 Mar;85(3):218-227. doi: 10.1037/ccp0000153. Epub 2016 Nov 3. PMID 27808536
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388
- [Derived] Tanofsky-Kraff M, Shomaker LB, Wilfley DE, Young JF, Sbrocco T, Stephens M, Ranzenhofer LM, Elliott C, Brady S, Radin RM, Vannucci A, Bryant EJ, Osborn R, Berger SS, Olsen C, Kozlosky M, Reynolds JC, Yanovski JA. Targeted prevention of excess weight gain and eating disorders in high-risk adolescent girls: a randomized controlled trial. Am J Clin Nutr. 2014 Oct;100(4):1010-8. doi: 10.3945/ajcn.114.092536. Epub 2014 Aug 13. PMID 25240070